CLINICAL TRIAL: NCT05380414
Title: A Single-center, Prospective Profiling Program of Advanced/Metastatic Pancreatic Cancer Patients
Brief Title: Profiling Program of Advanced/Metastatic Pancreatic Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ET21-399 GENOPANC
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Pancreatic Cancer; Advanced Pancreatic Cancer
Keywords: Molecular screening; Genomic profiles; Transcriptomic profiles
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic/advanced PDAC Patients (Experimental): Tumor samples
  Interventions: Biological: Tumor samples (archival FFPE) and blood samples

INTERVENTIONS:
Biological: Tumor samples (archival FFPE) and blood samples — Molecular screening

SUMMARY:
The proposal is to implement a molecular screening program for advanced/metastatic pancreatic cancer patients before the initiation of 1st line treatment in order to allow a better selection of patients for rationale personalized medicine with targeted agents and/or combination involving a chemotherapy backbone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient > 18 years
* metastatic or advanced PDAC
* Patient pretreated with no more than one prior systemic chemotherapy for metastatic/advanced disease (radiotherapy is not counted as a line of therapy).
* Availability of an archival representative FFPE tumor sample from primary tumor (surgery or diagnostic biopsy) and/or from metastatic lesion if metastatic disease at initial diagnosis with associated pathology report from an archival tumor block.
* Life expectancy > 3 months
* PS score 0 or 1.

Exclusion Criteria:

* Curative therapy available
* Any condition contraindicated with blood sampling procedures required by the protocol.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer.
* Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one actionable alteration defined as an alteration shown to predict for sensitivity to a drug FDA/EMA approved for use in another cancer type, or a relevant alteration for inclusion in a clinical trial. | At the end of study (5 years)

SECONDARY OUTCOMES:
Time from ICF signature to day 1 of next line of therapy | At day 1
Number of patients initiating a targeted therapy according to this molecular screening program with type of therapy initiated | At the end of study (5 years)
Progression-Free Survival (PFS) | Up to 12 months
Best overall response (BoR) | Up to 12 months
Overall survival (OS) | Up to 12 months
Duration of response (DoR) | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CASSIER, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France